CLINICAL TRIAL: NCT07258004
Title: OMNI Brain Health - An Investigation Into the Feasibility of Beetroot Juice Supplementation in People Living With Alzheimer's Disease.
Brief Title: An Investigation Into the Feasibility of Beetroot Juice Supplementation in People Living With Alzheimer's Disease.
Acronym: OMNI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of Scotland (Other)
Collaborators: NHS Lanarkshire (Other Government)
Responsible Party: Principal Investigator, Scott Nicol Findlay, Principal Investigator, University of the West of Scotland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OMNI Feasibility trial
Record Dates: First submitted 2025-11-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
Keywords: Nitric oxide; Dementia; Alzheimer's disease; Oral microbiome; Dietary nitrate; Beetroot juice
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beetroot juice supplementation (Experimental)
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Participants will take a concentrated beetroot juice shot (70ml) twice daily for 1-week. Each shot contains 400mg of dietary nitrate (800mg per day).

SUMMARY:
The goal of this clinical trial is to learn if taking a beetroot juice supplement will work in people living with Alzheimer's disease. The main questions it aims to answer are:

* Can people living with Alzheimer's disease realistically drink beetroot juice regularly (for example, is it easy to take, free from side effects and acceptable)?
* Does drinking beetroot juice twice a day improve health in people living with Alzheimer's disease?

Researchers will look at how you managed with the beetroot juice, as well as if there were any improvements in your health measures.

Participants will:

* Complete testing before and after the intervention for no more than 3 hours each time
* Complete a 1-day food diary before testing
* Take a beetroot juice supplementation twice daily for 1-week
* Keep a note of any problems with the beetroot juice

DETAILED DESCRIPTION:
Primary objectives:

To establish the feasibility of a beetroot juice supplement in people living with Alzheimer's disease (primary outcome). To establish whether a twice per day, 1-week beetroot juice intervention will induce changes in dementia related health outcomes (secondary outcomes).

Outline:

Participants will complete a 24-hour food diary prior to baseline testing before starting twice daily supplementation of beetroot juice shots for 7 days. Post-testing will be conducted on day 8 with a further 24-hour food diary having been completed prior to testing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-85 years
* Mild or Moderate Alzheimer's disease
* Participants must be able to speak, read, and understand English to participate in this study.
* To support adherence, participants are asked to have a carer, partner, friend, or family member available to assist with reminders to take the shots twice daily.

Exclusion Criteria:

* Advanced or severe Alzheimer's Disease
* Diagnosis of an additional neurological condition
* Have used antibiotics in the last month
* Use of mouthwash in the last month
* Use of medication affecting nitrate metabolism (for example proton pump inhibitors, Isosorbide Mononitrate, Sildenafil or Glyceryl Trinitrate).
* Unable to provide informed consent
* Allergies to beetroot
* Taking part in pharmacological trials

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a beetroot juice intervention in people living with Alzheimer's disease | From enrolment to the post-intervention testing 8-days later.
  Participants will be supported by a carer, friend or family member to complete a semi-structured interview to assess how feasible the trial was. Questions will be based around adherence (e.g. was the beetroot juice taken consistently and at the right times), acceptability/safety (e.g. was the beetroot juice tolerable and would they consider doing it daily if the benefits were proven and were there any adverse effects) and data collection feasibility (e.g. how easy was it to collect and post saliva samples themselves and how much of a burden was the pre and post-testing). Simple Likert scales will also be used to assess acceptability of the beetroot juice.

SECONDARY OUTCOMES:
Changes to oral microbiome pre to post intervention | From enrolment to the post-intervention testing 8-days later.
  An oral swab will collect bacteria from the tongue to analyse changes in the relative abundance of bacteria (%). Particular interest will be paid to pathogenic and nitrate reducing bacteria. Higher abundances of pathogenic bacteria and lower abundances of nitrate reducing bacteria indicate poorer oral health.
Changes to cognitive function pre and post intervention | From enrolment to the post-intervention testing 8-days later.
  Cognitive function will be assessed pre and post-intervention through the use of Montreal Cognitive Assessment. A different version of the questionnaire will be completed pre and post. Higher scores indicate better cognitive performance.
Changes to nitric oxide metabolism | From enrolment to the post-intervention testing 8-days later.
  Blood will be collected and analysed for arginine levels (µM). Higher nitric oxide levels can mean better health however, the inclusion of iNOS measurements is to determine the source of the nitric oxide i.e. whether it's inflammatory based, or health based.
Changes to nitric Oxide metabolism | From enrolment to the post-intervention testing 8-days later.
  Saliva and blood will be collected and analysed for nitric oxide levels (µM). Higher nitric oxide levels can mean better health however, the inclusion of iNOS measurements is to determine the source of the nitric oxide i.e. whether it's inflammatory based, or health based.
Changes to nitric oxide metabolism | From enrolment to the post-intervention testing 8-days later.
  Blood will be collected for arginase activity (µmol/min/mg protein). Higher arginase activity could mean better health however, the inclusion of iNOS measurements is to determine the source of the nitric oxide i.e. whether it's inflammatory based, or health based.
Changes to nitric oxide metabolism | From enrolment to the post-intervention testing 8-days later.
  Blood will be collected to analyse inducible nitric oxide synthase (iNOS) activity (relative fold change). Higher iNOS activity indicates greater levels of inflammation.
Changes in cardiovascular health pre to post intervention | From enrolment to the post-intervention testing 8-days later.
  Pulse wave analysis (augmentation index %) will be measured with lower scores considered better.
Change in body mass index pre to post intervention | From enrolment to the post-intervention testing 8-days later.
  Body mass index (kg/m²) will be calculated by measuring height (m) and weight (kg).
Changes in blood pressure pre to post intervention | From enrolment to the post-intervention testing 8-days later.
  Blood pressure (mmHg) will be measured with 120/80 considered normal.
Changes in exercise capacity pre to post intervention. | From enrolment to the post-intervention testing 8-days later.
  Exercise capacity will be measured with a 2-minute step in place test (more steps indicates a higher fitness level).
Changes in exercise levels pre to post intervention. | From enrolment to the post-intervention testing 8-days later.
  The International Physical Activity Questionnaire will be used to determine whether their physical activity levels change over the course of the intervention.
Changes to quality of life pre to post intervention. | From enrolment to the post-intervention testing 8-days later.
  Quality of life will be measured using Dementia Quality of Life questionnaire (DEMQOL). Higher scores indicate a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kimble, Study Director — University of the West of Scotland
Locations (1):
- University of the West of Scotland, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this feasibility trial will not be shared due to the small sample size and the sensitive nature of the data collected from participants with Alzheimer's disease. Sharing the data could risk participant re-identification and compromise privacy.